CLINICAL TRIAL: NCT03925584
Title: The Use of Music for Neonates Post-Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jean Connor, Director of Nursing Research, Cardiovascular and Critical Care Services, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00030729
Record Dates: First submitted 2019-03-15; First posted 2019-04-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: 1. To explore the feasibility of implementing standardized nurse-led music therapy for neonates post congenital heart surgery who are admitted to the cardiac intensive care unit.
  2. To describe the safety of implementing standardized nurse-led music therapy in the CICU.
  3. To gather data regarding sedation requirements of subjects during music therapy.
  4. To describe the parents perspective regarding nurse-led music therapy in the CICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy (Experimental): Implement standardized nurse-led music therapy for neonates post congenital heart surgery who are admitted to the cardiac intensive care unit.
  Interventions: Other: Music Therapy

INTERVENTIONS:
Other: Music Therapy — Standardized music playlist will be played centrally at the subjects head or feet for a period of 20 minutes once during a 12-hour shift for 14 days or until mechanical ventilation has been discontinued, whichever is first

SUMMARY:
The purpose of this study is to explore the feasibility of implementing nurse-led music therapy in a cohort of neonates admitted to the Cardiac Intensive Care Unit (CICU) post congenital heart surgery. In the proposed setting, the use of a standardized nurse-led music therapy protocol for post-operative neonates would build upon current successful nurse-led efforts to wean sedatives and opioid use for patients admitted to the CICU. The investigators believe data generated from this exploratory feasibility study may serve to further inform a larger study involving the use of music therapy in the cardiac intensive care.

DETAILED DESCRIPTION:
A predetermined recording of a music playlist meeting the properties of sedative music is being developed in consultation with a Boston Children's Hospital (BCH) music therapist. Properties of sedative music include soothing, stable, constant, and relatively unchanging, slow tempo and light rhythmic emphasis, constant volume and rhythm, lullaby style, repetitious and no separate melody for chorus/bridge. The music recorded for the neonates has been produced specifically for this study. In accordance with the recommendations for soothing music, BCH Music Therapists have recorded English nursery rhymes (Figure 1) in the key of C major at 60bpm with acoustic guitar and voice. The playlist will be stored on an Apple iPod Touch and will be delivered through a Bluetooth speaker that is positioned centrally (so that the sound input is received binaurally) at the subjects head or feet for a period of 20 minutes once during a 12-hour shift for 14 days or until mechanical ventilation has been discontinued, whichever is first.

The literature supports a duration of up to 30 minutes of music therapy followed by at least 30 minutes of silence, with a maximum of four hours per day. Music played for longer than 30 minutes has the potential to be a source of over-stimulation/agitation. There is some evidence to suggest that playing music for long periods of time (two four-hour segments) has a negative effect. In addition, it seems reasonable and likely to assume that the neonate could have a period of 30 minutes when they will not require an intervention associated with post-operative care. The protocol will target a 20 minute playlist. This will allow for variation in the length of songs while ensuring that music will not be played for longer than 30 minutes. There will be at least 30 minutes of quiet between music therapy session.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 37 weeks gestation,
* Between 0 to 30 days of age
* 24 hours post congenital heart surgery
* Receiving mechanical ventilation
* Background noise level (at bedside) at the time of music therapy must be 55dB or less.

Exclusion Criteria:

* Hemodynamically unstable or end of life
* If patient is in a closed Giraffe bed
* Evidence of hearing impairment
* Patient has known or suspected active seizure disorder

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of initiating music therapy protocol: Proportion of shifts with music therapy | 14 days or when mechanical ventilation is discontinued, whichever comes first
  Proportion of shifts with music therapy using the number of shifts during music therapy was initiated by number of eligible shifts
Feasibility of implementing 20-minute music therapy protocol: Proportion of shifts that the subject received the full 20- minute therapy uninterrupted | 14 days or when mechanical ventilation is discontinued, whichever comes first
  Proportion of shifts that the subject received the full 20- minute therapy uninterrupted using the number of shifts receiving the full therapy by the number of eligible therapy sessions

SECONDARY OUTCOMES:
Bedside nurse perception of music therapy | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  Bedside nurse will provide information on the ease or difficulty in administering the music therapy and to report any difficulties. Nurses will state if perceived the music therapy to provide any benefit as well as any additional comments or feedback.
Parent Satisfaction: survey | 24 hours following completion of music therapy
  Parents will be given a survey regarding satisfaction with the music therapy and any additional comments. Questions include satisfaction with music therapy, enjoyment of music, and beneficial/positive effects on infant and on parent themselves.
  Questions will be asked using a 5-point Likert scale ranging from Strongly Disagree to Strongly Agree. The rating for each question will range from 1 to 5. Strongly Disagree will be measured as 1, Disagree will be measured as 2, Neutral will be measured as 3, Agree will be measured as 4, and Strongly Agree will be measured as 5.
  The means/average of each question will be analysed. Questions rating 4.0 or higher will be considered as satisfaction. Average scores of 3.0-3.9 are considered Neutral, and Average scores below 3.0 are considered unsatisfied.
  There is also a section to allow for the parents to add additional comments on thoughts on the music therapy.
Physiological Measure - Heart Rate | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record the heart rate of the neonate.
Physiological Measure - Blood Pressure | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record the blood pressure (including systolic and diastolic pressures) of the neonate.
Physiological Measure - Oxygen Saturation | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record the oxygen saturation of the neonate.
Physiological Measure - State Behavioral Scale | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record the state behavioral scale (SBS) of the neonate. The SBS is determined by the Score as patient's response to voice then gentle touch then noxious stimuli (planned endotracheal suctioning or <5 seconds of nail bed pressure). SBS scores range from -3 to +2.
  The score for -3 is unresponsive, -2 is responsive to noxious stimuli, -1 is responsive to gentle touch or voice, 0 is awake and able to calm, +1 is restless and difficult to calm, and +2 is agitated.
Physiological Measure - Face, Legs, Activity, Cry, Consolability (FLACC) scale. | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record the FLACC scale of the neonate. Each category of the FLACC score is rated from 0 to 2. The total score ranges between 0 and 10.
  For Face, 0 is no particular expression or smile, 1 is occasional grimace or frown; withdrawn, disinterested, 2 is frequent to constant frown, clenched jaw, quivering chin.
  For Legs, 0 is normal position or relaxed, 1 is uneasy, restless, tense, 2 is kicking or legs drawn up.
  For Activity, 0 is lying quietly, normal position, moves easily, 1 is squirming, shifting back and forth, tense, 2 is arched, rigid, or jerking.
  For Cry, 0 is no cry (awake or asleep), 1 is moans or whimpers, occasional complaint, 2 is crying steadily, screams or sobs; frequent complaints.
  For Consolability, 0 is content, relaxed, 1 is reassured by occasional touching, hugging or being talked to; distractable, and 2 is difficult to console or comfort.
Measuring sedation | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record if sedation was given.
Music Frequency | Baseline and 5, 10, 20, 30, and 60 minutes from start of music therapy
  The beside nurses will record if the music therapy was stopped and the reason for stopping

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States